CLINICAL TRIAL: NCT03825341
Title: Hydroxyurea Therapy: Optimizing Access in Pediatric Populations Everywhere
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study terminated early due to challenges with recruitment during the COVID pandemic.
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HOPE18
Record Dates: First submitted 2019-01-23; First posted 2019-01-31 (Actual); Results first posted 2022-03-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-02

CONDITIONS: Sickle Cell Disease; Thalassemia
MeSH Terms: conditions — Anemia, Sickle Cell; Thalassemia | interventions — Hydroxyurea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 Liquid Hydroxyurea (Active Comparator): In Arm 1 of this study, n=18 infants ages 9 months to 2 years will be administered an extemporaneous oral liquid formulation of HU on a single occasion followed by PK sampling. The dose administered will be ~20 mg/kg/day or the infant's usual daily dose.
  Interventions: Drug: Hydroxyurea
- Arm 2 Hydroxyurea Oral Capsule (Active Comparator): In Arm 2, n=30 children who range in age from 2 to 18 years will be administered oral capsule HU, both a sprinkle formulation and capsules (Droxia® 200 mg), on two separate occasions separated by at least 1 but no more than 30 days in a randomized, crossover fashion. The doses of HU on each occasion will be rounded to the nearest 200 mg and will not exceed 35 mg/kg or 2000 mg
  Interventions: Drug: Hydroxyurea Oral Capsule

INTERVENTIONS:
Drug: Hydroxyurea — Drug: Hydroxyurea oral liquid dose administered will be 20mg/kg/day or infants's usual daily dose.
  Other Names: HU; Liquid Hydroxyurea
  Arms: Arm 1 Liquid Hydroxyurea
Drug: Hydroxyurea Oral Capsule — Drug: Hydroxyurea both a sprinkle formulation and capsules (Droxia 200mg) administered on 2 separate occasions.
  Other Names: HU Sprinkle; Doxroxia
  Arms: Arm 2 Hydroxyurea Oral Capsule

SUMMARY:
Primary Objective

1. Define the pharmacokinetics of liquid-formulated HU in infants (9 months to <2 years)
2. Assess the relative bioavailability of HU "sprinkles" compared to capsules in children and adolescents (≥2 to 18 years).

Secondary Objective:

Compare PK parameters in infants versus older children on this study and those from our previous "Pharmacokinetics and Bioavailability of a Liquid Formulation of Hydroxyurea in Pediatric Patients with Sickle Cell Anemia" (NCT01506544) trial.

Exploratory Objectives:

Capture information regarding the taste of HU sprinkles using palatability questionnaire.

This trial is an open label, single center assessment of the pharmacokinetics of two formulations of hydroxyurea (HU) designed to (1) determine the pharmacokinetic profile of a liquid formulation in infants and to (2) determine the bioavailability of "sprinkles", a novel method of administration for older children. The study aims to generate data to facilitate FDA approval for HU in children and potentially validate a new mode of administration ("sprinkles") that will optimize access and adherence for children in the US and globally.

DETAILED DESCRIPTION:
HOPE18 will be an open label, 2-arm study of HU disposition in 48 children with SCD. In Arm 1, n=18 infants ages 9 months to 2 years will be administered an extemporaneous oral liquid formulation of HU on a single occasion followed by PK sampling. The dose administered will be ~20 mg/kg/day or the infant's usual daily dose. In Arm 2, n=30 children who range in age from 2 to 18 years will be administered HU, both a sprinkle formulation and capsules (Droxia® 200 mg), on two separate occasions separated by at least 1 day but no more than 30 days in a randomized, crossover fashion. The doses of HU on each occasion will be rounded to the nearest 200 mg and will not exceed 35 mg/kg or 2000 mg. We hypothesize that the PK profile of the sprinkle formulation will not differ significantly from the PK profile of Droxia® capsules in children and adolescents ages ≥2 - 18 years of age. Participants in both arms will be followed up to 30 days from receiving last HU dose.

ELIGIBILITY:
Inclusion Criteria:

Participants will be eligible for this study if only if all of the following inclusion criteria apply:

* Laboratory (i.e. electrophoretic, chromatographic or DNA) confirmation of HbSS or HbSβ0thalassemia.
* Participants may or may not be currently receiving HU. If participants are taking HU, then their most recent dose must be ≥24 hours prior to the start of the study.
* Participant is in the "well" state (defined by ≥ 2 weeks since the last SCD-related complication).
* Clinical evidence of normal gastrointestinal function and structure.
* No clinical evidence of hepatic compromise, including transaminases < 3 times the upper limit of normal.
* Estimated glomerular filtration rate (Schwartz equation) > 70 ml/min/1.73m2.
* Body mass index (BMI) ≥5th and ≤95th percentile as per CDC growth charts.

In addition:

For the Pharmacokinetic Study (Arm 1):

* Age ≥ 9 months and < 2 years.
* Able to consume a minimum of 30 ml of water following ingestion of the study article.

For the Bioavailability Study (Arm 2):

* Age ≥ 2 years and ≤ 18 years.
* Weight of ≥ 10 kg
* Females of child-bearing potential must have a negative pregnancy test prior to dosing and be willing to practice appropriate contraceptive measures, including abstinence, from the time of the initial pregnancy testing through the remainder of the study (30 days after last administration of investigational agents).
* Males of child-bearing potential must be willing to practice appropriate contraceptive measures, including abstinence, during study participation (30 days after last administration of investigational agents).
* Able to ingest both sprinkles and capsule study articles and consume a minimum of 30 ml of water following ingestion of each agent.

Exclusion Criteria:

* Chronic transfusion therapy, or transfused within 3 months of study participation.
* Known renal impairment (creatinine >1.5x the upper limit of normal for age).
* Known hepatic impairment or Grade 2 or higher transaminases and bilirubin levels.
* Diagnoses other than sickle cell anemia or sickle beta-zero thalassemia (i.e., other sickle cell variants or sickle/ hereditary persistence of fetal hemoglobin).
* Blood count parameters as follows: hemoglobin <6.0 gm/dL, absolute reticulocyte count <80,000/mm3, absolute neutrophil count <1000/mm3, or platelet count <80,000/mm3.
* The participant has used opiates, H2 blockers, proton pump inhibitors, antacids, other GI motility agents or any other medication that, in the opinion of the investigator, will interfere with the study procedures or affect the interpretation of the results of the study for 3 days prior to the first dose of study.
* Participants taking antiretroviral drugs (including didanosine and stavudine) due to increased risk of toxicity with concomitant use.
* Participation in another clinical intervention trial utilizing an IND/IDE agent, but can participate in HUGKISS since same drug agent.

Ages: 9 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremie Estepp, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1 participant was recruited between March 2019 and Jan. 2022. The participant was randomized but did not receive treatment.
Period: Overall Study
Arm/Group | Arm 1 Liquid Hydroxyurea | Arm 2 Hydroxyurea Oral Capsule
Started | 0 | 1
Completed | 0 | 0
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: No enrollments on Arm 1.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 Liquid Hydroxyurea | Arm 2 Hydroxyurea Oral Capsule | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Categorical [Count of Participants; unit: Participants] — Population: Baseline data not entered for the 1 enrollment due to confidentiality concerns.
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Baseline data not entered for the 1 enrollment due to confidentiality concerns.
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Baseline data not entered for the 1 enrollment due to confidentiality concerns.
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Baseline data not entered for the 1 enrollment due to confidentiality concerns.

OUTCOME MEASURES:

1. Primary Outcome: The Maximum Concentration Observed After Dosing (Cmax) for HU Liquid Formulation in Infants (9 Months to <2 Years)
Description: Summary statistics including mean, standard deviation (SD) will be reported.
Time Frame: 1 day
Population: No participants were enrolled on Arm 1.
Arm/Group | Arm 1 Liquid Hydroxyurea
Number analyzed (Participants) | 0

2. Primary Outcome: The Time of Maximum Observed Concentration (Cmax) Relative to Time of Dosing for HU Liquid Formulation in Infants (9 Months to <2 Years)
Description: Summary statistics including mean, standard deviation (SD) will be reported.
Time Frame: 1 day
Population: No participants were enrolled on Arm 1.
Arm/Group | Arm 1 Liquid Hydroxyurea
Number analyzed (Participants) | 0

3. Primary Outcome: AUClast for HU Liquid Formulation in Infants (9 Months to <2 Years)
Description: The area under the concentration-time curve from time of dosing of the drug to the time of the last measurable concentration or when concentrations were Below the Limit of Quantitation (BLQ) were calculated using either the linear (concentration before Cmax) or log trapezoidal rule (concentrations after Cmax). Summary statistics including mean, standard deviation (SD) will be reported.
Time Frame: 1 day
Population: No participants were enrolled on Arm 1.
Arm/Group | Arm 1 Liquid Hydroxyurea
Number analyzed (Participants) | 0

4. Primary Outcome: AUCinfinity for HU Liquid Formulation in Infants (9 Months to <2 Years)
Description: The AUC extrapolated from the last measured concentration (Clast) to time infinity using the formula AUClast + Clast / λz. Summary statistics including mean, standard deviation (SD) will be reported.
Time Frame: 1 day
Population: No participants were enrolled on Arm 1.
Arm/Group | Arm 1 Liquid Hydroxyurea
Number analyzed (Participants) | 0

5. Primary Outcome: Mean Residence Time as Generated by WinNonlin (AUMC/AUC) for HU Liquid Formulation in Infants (9 Months to <2 Years)
Description: Summary statistics including mean, standard deviation (SD) will be reported.
Time Frame: 1 day
Population: No participants were enrolled on Arm 1.
Arm/Group | Arm 1 Liquid Hydroxyurea
Number analyzed (Participants) | 0

6. Primary Outcome: Apparent Clearance Calculated From Dose/ AUCINF for HU Liquid Formulation in Infants (9 Months to <2 Years)
Description: Summary statistics including mean, standard deviation (SD) will be reported.
Time Frame: 1 day
Population: No participants were enrolled on Arm 1.
Arm/Group | Arm 1 Liquid Hydroxyurea
Number analyzed (Participants) | 0

7. Primary Outcome: Apparent Clearance Normalized for Body Weight (BW) for HU Liquid Formulation in Infants (9 Months to <2 Years)
Description: Summary statistics including mean, standard deviation (SD) will be reported.
Time Frame: 1 day
Population: No participants were enrolled on Arm 1.
Arm/Group | Arm 1 Liquid Hydroxyurea
Number analyzed (Participants) | 0

8. Primary Outcome: Elimination Slope for HU Liquid Formulation in Infants (9 Months to <2 Years)
Description: The first-order linear slope associated with the terminal (log-linear) portion of the curve and estimated via linear regression of log concentrations vs. time. Summary statistics including mean, standard deviation (SD) will be reported.
Time Frame: 1 day
Population: No participants were enrolled on Arm 1.
Arm/Group | Arm 1 Liquid Hydroxyurea
Number analyzed (Participants) | 0

9. Primary Outcome: Terminal Elimination Half-life Obtained From: t½ = ln(2)/ λz for HU Liquid Formulation in Infants (9 Months to <2 Years)
Description: Summary statistics including mean, standard deviation (SD) will be reported.
Time Frame: 1 day
Population: No participants were enrolled on Arm 1.
Arm/Group | Arm 1 Liquid Hydroxyurea
Number analyzed (Participants) | 0

10. Secondary Outcome: The Maximum Concentration Observed After Dosing (Cmax) for HU "Sprinkles" Compared to Capsules in Children and Adolescents (≥2 to 18 Years)
Description: Summary statistics including mean and SD will be reported for "sprinkles" and capsules and will be compared using two-sample t-test or Wilcoxon rank sum test depending on the normality of the data at a significance level of 0.05 per study design above. Logarithmic transformation will be applied if data do not follow normal.
Time Frame: 2 days
Population: No participants treated on Arm 2.
Arm/Group | Arm 2 Hydroxyurea Oral Capsule
Number analyzed (Participants) | 0

11. Secondary Outcome: The Time of Maximum Observed Concentration (Cmax) Relative to Time of Dosing for HU "Sprinkles" Compared to Capsules in Children and Adolescents (≥2 to 18 Years)
Description: as for outcome 10
Time Frame: 2 days
Population: No participants treated on Arm 2.
Arm/Group | Arm 2 Hydroxyurea Oral Capsule
Number analyzed (Participants) | 0

12. Secondary Outcome: AUClast for HU "Sprinkles" Compared to Capsules in Children and Adolescents (≥2 to 18 Years)
Description: The AUC extrapolated from the last measured concentration (Clast) to time infinity using the formula AUClast + Clast / λz. Summary statistics including mean and SD will be reported for "sprinkles" and capsules and will be compared using two-sample t-test or Wilcoxon rank sum test depending on the normality of the data at a significance level of 0.05 per study design above. Logarithmic transformation will be applied if data do not follow normal.
Time Frame: 2 days
Population: No participants treated on Arm 2.
Arm/Group | Arm 2 Hydroxyurea Oral Capsule
Number analyzed (Participants) | 0

13. Secondary Outcome: AUCinfinity for HU "Sprinkles" Compared to Capsules in Children and Adolescents (≥2 to 18 Years)
Description: as for outcome 12
Time Frame: 2 days
Population: No participants treated on Arm 2.
Arm/Group | Arm 2 Hydroxyurea Oral Capsule
Number analyzed (Participants) | 0

14. Secondary Outcome: Mean Residence Time as Generated by WinNonlin (AUMC/AUC) for HU "Sprinkles" Compared to Capsules in Children and Adolescents (≥2 to 18 Years)
Description: as for outcome 10
Time Frame: 2 days
Population: No participants treated on Arm 2.
Arm/Group | Arm 2 Hydroxyurea Oral Capsule
Number analyzed (Participants) | 0

15. Secondary Outcome: Apparent Clearance Calculated From Dose/ AUCINF for HU "Sprinkles" Compared to Capsules in Children and Adolescents (≥2 to 18 Years)
Description: as for outcome 10
Time Frame: 2 days
Population: No participants treated on Arm 2.
Arm/Group | Arm 2 Hydroxyurea Oral Capsule
Number analyzed (Participants) | 0

16. Secondary Outcome: Apparent Clearance Normalized for Body Weight (BW) for HU "Sprinkles" Compared to Capsules in Children and Adolescents (≥2 to 18 Years)
Description: as for outcome 10
Time Frame: 2 days
Population: No participants treated on Arm 2.
Arm/Group | Arm 2 Hydroxyurea Oral Capsule
Number analyzed (Participants) | 0

17. Secondary Outcome: Elimination Slope for HU "Sprinkles" Compared to Capsules in Children and Adolescents (≥2 to 18 Years)
Description: The first-order linear slope associated with the terminal (log-linear) portion of the curve and estimated via linear regression of log concentrations vs. time. Summary statistics including mean and SD will be reported for "sprinkles" and capsules and will be compared using two-sample t-test or Wilcoxon rank sum test depending on the normality of the data at a significance level of 0.05 per study design above. Logarithmic transformation will be applied if data do not follow normal.
Time Frame: 2 days
Population: No participants treated on Arm 2.
Arm/Group | Arm 2 Hydroxyurea Oral Capsule
Number analyzed (Participants) | 0

18. Secondary Outcome: Terminal Elimination Half-life Obtained From: t½ = ln(2)/ λz for HU "Sprinkles" Compared to Capsules in Children and Adolescents (≥2 to 18 Years)
Description: as for outcome 10
Time Frame: 2 days
Population: No participants treated on Arm 2.
Arm/Group | Arm 2 Hydroxyurea Oral Capsule
Number analyzed (Participants) | 0

19. Secondary Outcome: The Maximum Concentration Observed After Dosing (Cmax) for Infants Versus Older Children
Description: The older children will include children on arm 2 on this study and those from our previous "Pharmacokinetics and Bioavailability of a Liquid Formulation of Hydroxyurea in Pediatric Patients with Sickle Cell Anemia" (NCT01506544) trial. Summary statistics will be reported for the infants and older children and will be compared using two sample t-test or Wilcoxon rank sum test depending on the normality of the data. Logarithmic transformation will be applied if data do not follow normal.
Time Frame: 2 days
Population: No participants were treated on this study.
Arm/Group | Arm 1 Liquid Hydroxyurea | Arm 2 Hydroxyurea Oral Capsule
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: The Time of Maximum Observed Concentration (Cmax) Relative to Time of Dosing for Infants Versus Older Children
Description: as for outcome 19
Time Frame: 2 days
Population: No participants were treated on this study.
Arm/Group | Arm 1 Liquid Hydroxyurea | Arm 2 Hydroxyurea Oral Capsule
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: AUClast for Infants Versus Older Children
Description: The area under the concentration-time curve from time of dosing of the drug to the time of the last measurable concentration or when concentrations were Below the Limit of Quantitation (BLQ) were calculated using either the linear (concentration before Cmax) or log trapezoidal rule (concentrations after Cmax). The older children will include children on arm 2 on this study and those from our previous "Pharmacokinetics and Bioavailability of a Liquid Formulation of Hydroxyurea in Pediatric Patients with Sickle Cell Anemia" (NCT01506544) trial. Summary statistics will be reported for the infants and older children and will be compared using two sample t-test or Wilcoxon rank sum test depending on the normality of the data. Logarithmic transformation will be applied if data do not follow normal.
Time Frame: 2 days
Population: No participants were treated on this study.
Arm/Group | Arm 1 Liquid Hydroxyurea | Arm 2 Hydroxyurea Oral Capsule
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: AUCinfinity for Infants Versus Older Children
Description: The AUC extrapolated from the last measured concentration (Clast) to time infinity using the formula AUClast + Clast / λz. The older children will include children on arm 2 on this study and those from our previous "Pharmacokinetics and Bioavailability of a Liquid Formulation of Hydroxyurea in Pediatric Patients with Sickle Cell Anemia" (NCT01506544) trial. Summary statistics will be reported for the infants and older children and will be compared using two sample t-test or Wilcoxon rank sum test depending on the normality of the data. Logarithmic transformation will be applied if data do not follow normal.
Time Frame: 2 days
Population: No participants were treated on this study.
Arm/Group | Arm 1 Liquid Hydroxyurea | Arm 2 Hydroxyurea Oral Capsule
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Mean Residence Time as Generated by WinNonlin (AUMC/AUC) for Infants Versus Older Children
Description: as for outcome 19
Time Frame: 2 days
Population: No participants were treated on this study.
Arm/Group | Arm 1 Liquid Hydroxyurea | Arm 2 Hydroxyurea Oral Capsule
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: Apparent Clearance Calculated From Dose/ AUCINF for In Infants Versus Older Children
Description: as for outcome 19
Time Frame: 2 days
Population: No participants were treated on this study.
Arm/Group | Arm 1 Liquid Hydroxyurea | Arm 2 Hydroxyurea Oral Capsule
Number analyzed (Participants) | 0 | 0

25. Secondary Outcome: Apparent Clearance Normalized for Body Weight (BW) for Infants Versus Older Children
Description: as for outcome 19
Time Frame: 2 days
Population: No participants were treated on this study.
Arm/Group | Arm 1 Liquid Hydroxyurea | Arm 2 Hydroxyurea Oral Capsule
Number analyzed (Participants) | 0 | 0

26. Secondary Outcome: Elimination Slope for In Infants Versus Older Children
Description: The first-order linear slope associated with the terminal (log-linear) portion of the curve and estimated via linear regression of log concentrations vs. time. The older children will include children on arm 2 on this study and those from our previous "Pharmacokinetics and Bioavailability of a Liquid Formulation of Hydroxyurea in Pediatric Patients with Sickle Cell Anemia" (NCT01506544) trial. Summary statistics will be reported for the infants and older children and will be compared using two sample t-test or Wilcoxon rank sum test depending on the normality of the data. Logarithmic transformation will be applied if data do not follow normal.
Time Frame: 2 days
Population: No participants were treated on this study.
Arm/Group | Arm 1 Liquid Hydroxyurea | Arm 2 Hydroxyurea Oral Capsule
Number analyzed (Participants) | 0 | 0

27. Secondary Outcome: Terminal Elimination Half-life Obtained From: t½ = ln(2)/ λz for Infants Versus Older Children
Description: as for outcome 19
Time Frame: 2 days
Population: No participants were treated on this study.
Arm/Group | Arm 1 Liquid Hydroxyurea | Arm 2 Hydroxyurea Oral Capsule
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: No participants were treated on this study.
Description: No participants were treated on this study.
Arm/Group | Arm 1 Liquid Hydroxyurea | Arm 2 Hydroxyurea Oral Capsule
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
No participants were treated on this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-03-26): https://cdn.clinicaltrials.gov/large-docs/41/NCT03825341/Prot_SAP_000.pdf
  • Informed Consent Form (2018-12-21): https://cdn.clinicaltrials.gov/large-docs/41/NCT03825341/ICF_001.pdf